CLINICAL TRIAL: NCT02773615
Title: CT Perfusion Added to CT Angiography for Unstable Angina or Nonanginal Chest Pain in the Emergency Department (PERFeCT) : a Feasibility and Safety Pilot Study.
Brief Title: CT Perfusion Added to CT Angiography
Acronym: PERFeCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, dr. Kaatje Goetschalckx, Dr in Cardiovascular Medicine, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S59077
Record Dates: First submitted 2016-05-03; First posted 2016-05-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac computed tomography — Non-invasive CT scan of the heart

SUMMARY:
Background In the differential diagnosis of unstable angina versus non-anginal chest pain, an exercise test is often the modality of choice for further investigation. However, in a substantial number of patients exercise testing is less informative, because of insufficient exercise capacity or pre-existing ECG-abnormalities. In patients with low pretest probability of coronary artery disease (CAD), Coronary CT angiography (CTA) has an excellent negative predictive value, but in patients with an intermediate or high pretest probability of CAD estimation of the hemodynamic significance of a stenosis has only limited specificity. CT perfusion (CTP) is a new method looking at myocardial perfusion during vasodilative stress with a sensitivity, specificity, positive predictive value and negative predictive value of respectively 81%, 93%, 87% and 88%, whereas radiation is limited to a maximum of 5 millisievert (mSv).

Aim It is the aim of this pilot study to investigate whether the addition of CTP to CTA is a feasible and safe investigational workflow in patients with unstable angina or nonanginal chest pain in the emergency department.

DETAILED DESCRIPTION:
It is the aim of this pilot study to investigate whether the addition of CTP to CTA is a feasible and safe investigational workflow in patients with unstable angina or nonanginal chest pain in the emergency department.

Methods Patients presenting in the emergency department with thoracic pain or other symptoms suggestive of angina, will be eligible for the study if there are no ECG-signs of acute ischemia (no STEMI or NSTEMI) and if 2 serial high sensitivity Troponin T measurements with an interval of 1 hour are not conclusive for the diagnosis of ischemia.

Exclusion criteria are a history of a STEMI or a NSTEMI with residual functional abnormalities, atrial fibrillation, renal insufficiency with glomerular filtration rate (GFR) < 60 ml/min or known contrast allergy. A number of 100 patients in one year is targeted.

A pretest-probability score is calculated based on age, gender and type of angina of the patient. Typical angina is defined as substernal chest pain or discomfort provoked by exertion or emotional stress and relieved by rest or nitrates within minutes, atypical angina meets 2 of the 3 characteristics and nonanginal pain meets one or none of the characteristics. The time point of admission in the emergency department is recorded.(cf. Figure 1) Patients will undergo a CT (Siemens Somatom Force) with calcium-scoring and CT angiography (CTA). The amount of contrast used is about 60 ml, and the radiation varies between 0.5 and 1.5 mSv. If the CTA is completely normal and Ca-scoring is low (< 100), no further investigations are performed and the diagnosis of nonanginal pain is probable. Patients are dismissed from the emergency ward with follow-up organized for one year. Cf. Figure 2.

If there are abnormalities on CTA, or if there is a elevated Ca-scoring (> 300), even in the absence of stenosis on CTA, a CT perfusion sequence is added during dipyridamole stress. The amount of contrast used for CTP is about 50 ml and the radiation used for CTP varies between 3 to 4 mSv, resulting in a total radiation dose of less than 5 mSv. Dipyridamole is administered in a dose of 140 µg/kg body weight/minute during 6 minutes through a peripheral vein. CTP is performed 2 minutes after completion of the dipyridamole infusion.

If CTP is suggestive of cardiac ischemia, defined as a visual perfusion defect, an invasive coronary angiography, with fractional flow measurement if needed, will be performed.

If CTP is negative, defined as no visual perfusion defect, no further investigations are performed and the diagnosis of nonanginal pain is probable. Patients are dismissed from the emergency ward with follow-up for one year. Cf. Figure 2.

At dismissal, patients are asked to fill in an angina-questionnaire (short form Seattle Angina Questionnaire, SAQ) , a quality of life (SF-12 Health Survey) , and a satisfaction questionnaire about the hospital stay and investigational flow). The time point of dismissal is recorded.

After dismissal, patients are contacted after 3 months to ask for hospitalizations or investigations that might have occurred in the mean time, and to fill in the same SAQ and SF-12. At 12 months after the initial presentation, patients are invited to a cardiac consultation and questionnaires are completed for the last time.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with chest pain in the ED
* ≥ 18 years of age
* Patient is stable and in adequate clinical condition to undergo CTA + CTP

Exclusion Criteria:

* no ECG-signs of acute ischemia (no STEMI or NSTEMI)
* Hs Troponine T level/evolution indicative of ischemia
* history of a STEMI or a NSTEMI with residual functional abnormalities
* atrial fibrillation
* renal insufficiency with glomerular filtration rate (GFR) =< 30 ml/min
* Hb < 8.5 g/dL
* Infection with systemic involvement
* Baseline respiratory failure requiring oxygen at home
* Severe COPD
* Intrinsic astma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting in the emergency department with thoracic pain or other symptoms suggestive of angina, will be eligible for the study if there are no ECG-signs of acute ischemia (no STEMI or NSTEMI) and if 2 serial high sensitivity Troponine T measurements with an interval of 1 hour are not conclusive for the diagnosis of ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival | two years
  Registration of adverse cardiac events during clinical follow up

SECONDARY OUTCOMES:
Quality of life | two years
  Assessment of quality of life using the Seattle Angina Questionnaire (SAQ7)
Quality of life second | two years
  Quality-of-life (SF-12 health survey) questionnaire.
Impact of CTP on the diagnostic accuracy for the detection of obstructive CAD | two years
  Evaluated according to pre test probability

CONTACTS AND LOCATIONS:
Overall Officials: Kaatje Goetschalckx, MD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Athanasiadis A, Sechtem U; European Society of Cardiology. [Diagnostics and therapy of chronic stable coronary artery disease : new guidelines of the European Society of Cardiology]. Herz. 2014 Dec;39(8):902-12. doi: 10.1007/s00059-014-4159-1. German. PMID 25384852
- [Background] Williams MC, Newby DE. CT myocardial perfusion imaging: current status and future directions. Clin Radiol. 2016 Aug;71(8):739-49. doi: 10.1016/j.crad.2016.03.006. Epub 2016 Apr 16. PMID 27091433